CLINICAL TRIAL: NCT03468985
Title: A Randomized Phase II Trial of Nivolumab, Cabozantinib Plus Nivolumab, and Cabozantinib Plus Nivolumab Plus Ipilimumab in Patients With Previously Treated Non-Squamous NSCLC
Brief Title: Nivolumab, Cabozantinib S-Malate, and Ipilimumab in Treating Patients With Recurrent Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01008; NCI-2017-01008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5152 (Other: ECOG-ACRIN Cancer Research Group); EA5152 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Lung Non-Squamous Non-Small Cell Carcinoma; Recurrent Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
Keywords: Nivolumab; Cabozantinib; Ipilimumab; NSCLC
MeSH Terms: interventions — cabozantinib; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (nivolumab) (Active Comparator): Patients receive nivolumab IV over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab
- Arm B (nivolumab, cabozantinib) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1 and cabozantinib s-malate PO daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Biological: Nivolumab
- Arm C (nivolumab, cabozantinib, ipilimumab) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1, cabozantinib s-malate PO daily on days 1-28, and ipilimumab IV over 90 minutes every 8 weeks. Cycles for nivolumab and cabozantinib s-malate repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Biological: Ipilimumab; Biological: Nivolumab
- Arm T (Targeted cohort; nivolumab, cabozantinib) (Experimental): Patients with ROS1 gene rearrangement, MET exon 14 splice mutations, MET high amplification, or RET gene rearrangement receive nivolumab IV over 60 minutes on day 1 and cabozantinib s-malate PO daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Biological: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Given PO
  Other Names: Cabozantinib s-malate; XL-184; EXEL-7184; EXEL-02977184; Cabometyx®
  Arms: Arm B (nivolumab, cabozantinib); Arm C (nivolumab, cabozantinib, ipilimumab); Arm T (Targeted cohort; nivolumab, cabozantinib)
Biological: Ipilimumab — Given IV
  Other Names: Anti-CTLA-4 monoclonal antibody; MDX-010; Yervoy
  Arms: Arm C (nivolumab, cabozantinib, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX1106

SUMMARY:
This partially randomized phase II trial studies how well nivolumab, cabozantinib s-malate, and ipilimumab work in treating patients with stage IV non-small cell lung cancer that has come back. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving nivolumab, cabozantinib s-malate, and ipilimumab may work better than cabozantinib s-malate alone in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate whether combination therapy of nivolumab and cabozantinib s-malate (cabozantinib), or of nivolumab and cabozantinib, and ipilimumab as compared to nivolumab alone, extends progression-free survival (PFS) for this patient population with non-squamous non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To estimate the overall survival for each arm of the trial. II. To estimate the best overall response rate for each arm of the trial. III. To estimate the progression free survival of the targeted therapy arm of the trial.

IV. To describe the toxicity profile of monotherapy with nivolumab, and the combination of nivolumab and cabozantinib, and the combination of nivolumab and cabozantinib and ipilimumab, in this patient population with non-squamous NSCLC.

CORRELATIVE OBJECTIVES:

I. To adjust progression free survival for each arm based on PD-L1 tumor status.

IMAGING OBJECTIVES:

I. To describe time point tumor response assessment, overall best response and progression-free survival using the conventional Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and the exploratory uni-dimensional immune response criteria (iRRC) and the imaging (i)RECIST criteria with all measurements performed by the central review.

II. To compare RECIST 1.1 imaging response assessment measurements (time point response assessment and overall best response) assess by site study personnel to those performed by central review.

EXPLORATORY TOBACCO USE OBJECTIVES:

I. To determine the effects of tobacco, operationalized as combustible tobacco (1a), other forms of tobacco (1b), and environmental tobacco exposure (ETS) (1c) on provider-reported cancer-treatment toxicity (adverse events (both clinical and hematologic) and dose modifications).

II. To determine the effects of tobacco on patient-reported physical symptoms and psychological symptoms.

III. To examine quitting behaviors and behavioral counseling/support and cessation medication utilization.

IV. To explore the effect of tobacco use and exposure on treatment duration, relative dose intensity, and therapeutic benefit.

OUTLINE: Patients are randomized to 1 of 3 arms. Patients with ROS1 gene rearrangement, MET exon 14 splice mutations, MET high amplification, or RET gene rearrangement are assigned to Arm T.

ARM A: Patients receive nivolumab at 480 mg intravenously (IV) over 60 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive nivolumab at 480 mg IV over 60 minutes on day 1 and cabozantinib s-malate at 40 mg orally (PO) daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive nivolumab at 480 mg IV over 60 minutes on day 1, cabozantinib s-malate at 40 mg PO daily on days 1-28, and ipilimumab at 1 mg/kg IV over 90 minutes every 8 weeks. Cycles for nivolumab and cabozantinib s-malate repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM T: Patients with ROS1 gene rearrangement, MET exon 14 splice mutations, MET high amplification, or RET gene rearrangement receive nivolumab at 480 mg IV over 60 minutes on day 1 and cabozantinib s-malate at 40 mg PO daily on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria (Step 0):

* Patients with tumors with the following molecular alterations must submit testing results via Medidata Rave to determine eligibility to Arm T; the study chair, co-chair, biology co-chair, or a delegate must review the molecular testing and agree that the testing meets one of the molecular eligibility criteria below:

  * ROS1 gene rearrangement by fluorescence in situ hybridization (FISH) or deoxyribonucleic acid (DNA) analysis (may have progressed on prior crizotinib therapy)
  * MET exon 14 splice mutations on DNA analysis (may have progressed on prior crizotinib therapy)
  * MET high amplification by FISH or DNA analysis or other MET mutations predicted to be sensitive to MET inhibitor (no prior targeted therapy allowed)
  * RET gene rearrangement by FISH or DNA analysis (no prior targeted therapy allowed)

    * Institutions will be notified of the patient's eligibility status for Arm T within two (2) business days of submission of the molecular testing reports
    * If patients do not have tumors with the above molecular alterations noted proceed directly to step 1

Inclusion Criteria (Step 1):

* For patients with known molecular alterations, institution has been notified that patient is deemed eligible for Arm T per review of molecular testing reports
* Pathologically confirmed non-squamous non-small cell lung carcinoma (NSCLC)
* Stage IV disease (includes M1a, M1b, or recurrent disease), according to the 7th edition of the lung cancer tumor, node, and metastasis (TNM) classification system
* Predominant non-squamous histology (patients with NSCLC not otherwise specified [NOS] are eligible); mixed tumors will be categorized by the predominant cell type; if small cell elements are present the patient is ineligible
* Tumors must be tested and known negative for EGFR tyrosine kinase inhibitor (TKI) sensitizing mutations (EGFR exon 19 deletions, L858R, L861Q, G719X) and ALK gene rearrangements by routine Clinical Laboratory Improvement Act (CLIA)-certified clinical testing methods; negative circulating tumor DNA results alone are not acceptable; prior testing for tumor PD-L1 status is not required
* Patients must have progressed radiographically following first line platinum-based chemotherapy, no additional lines of therapy are permitted

  * NOTE: Prior adjuvant chemotherapy for early stage disease does not count as one line of therapy if 12 months or greater elapsed between completion of adjuvant therapy and initiation of first-line systemic therapy; if less than 12 months elapsed, adjuvant chemotherapy counts as one line of therapy
  * Exception for targeted therapy sub-study (Arm T): At least one line of prior chemotherapy or targeted therapy is required, but there is no limit on number of prior treatments
* Patients must have measurable disease as defined by RECIST v. 1.1 criteria; baseline measurements and evaluation of all sites of disease must be obtained within 4 weeks prior to registration
* Any prior chemotherapy (based on administration schedule) must have been completed in greater than or equal to the following times prior to registration:

  * Chemotherapy/ targeted oral therapy administered in a daily or weekly schedule must be completed >= 1 week prior to registration;
  * Any chemotherapy administered in an every 2 week or greater schedule must be completed >= 2 weeks prior to registration
  * Additionally, patients should be recovered to equal to or less than grade 1 toxicities related to any prior treatment, unless adverse event (AE)(s) are clinically nonsignificant and/or stable on supportive therapy
* Patients with no known brain metastasis must have baseline brain imaging within 12 weeks prior to study registration not demonstrating brain metastases OR patients with known brain metastases must have baseline brain imaging within 4 weeks prior to study registration and meet all of the following criteria:

  * Have completed treatment to all symptomatic brain metastases (with whole brain radiation or radiosurgery) >= 4 weeks prior to registration, or have undergone complete neurosurgical resection >= 3 months prior to registration
  * Be clinically stable from brain metastases at time of screening, if no treatment was administered
  * Known leptomeningeal disease is not allowed
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have anticipated life expectancy greater than 3 months
* Absolute neutrophil count >= 1,500/mm^3 (within 2 weeks prior to registration)
* Platelets >= 100,000/mm^3 (within 2 weeks prior to registration)
* Hemoglobin >= 9 g/dL (within 2 weeks prior to registration)
* Subject has prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) test =< 1.3 x the laboratory upper limit of normal (ULN) (within 2 weeks prior to registration)
* Total bilirubin =< 1.5 x ULN (within 2 weeks prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN (within 2 weeks prior to registration)
* Serum albumin >= 2.8 g/dL (within 2 weeks prior to registration)
* Serum calcium (absolute or albumin corrected), magnesium and potassium >= lower limit of normal (LLN) (within 2 weeks prior to registration)

  * NOTE: serum calcium, magnesium and potassium can be replaced if values are below LLN
* Creatinine =< 1.5 x ULN or calculated (Cockcroft-Gault formula) or measured creatinine clearance >= 50 mL/min/1.73 m^2 (normalized to body surface area [BSA]) for patients with creatinine levels greater than 1.5 times the institutional normal (within 2 weeks prior to registration)
* Screening urine dipstick must equal 0 or "trace"; if urine dipstick results are >= 1+, or if dipstick was not performed, calculation of urine protein creatinine (UPC) is required and patients must have a UPC ratio =< 1 to participate in the study (within 2 weeks prior to registration)
* Patients must have corrected QT interval calculated by the Fridericia formula (QTcF) =< 500 ms within 28 days before registration
* Patients must be able to swallow tablets

  * All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential (WOCBP) and males who are sexually active with WOCBP must use an accepted and effective method of contraception or abstain from sexual intercourse for at least one week prior to the start of treatment, and continue for 5 months after the last dose of protocol treatment for women of childbearing potential and 7 months after the last dose of protocol treatment for males who are sexually active with WOCBP

Exclusion Criteria (Step 1):

* Small cell elements are present
* Prior anti-MET therapy such as crizotinib or cabozantinib, or PD-1/PD-L1 immune checkpoint inhibitor therapy (such as nivolumab, pembrolizumab, atezolizumab) or CTLA4 inhibitor therapy (such as ipilimumab); prior allergic reaction to small molecule tyrosine kinase inhibitors or monoclonal antibodies

  * Exception for targeted therapy sub-study (Arm T): Prior crizotinib may be allowed depending on the gene alteration
* Prior radiation therapy for bone metastasis within 2 weeks; any other radiation therapy within 4 weeks prior to registration
* Known leptomeningeal disease
* Impaired decision-making capacity (IDMC)
* Clinically-significant gastrointestinal bleeding within 6 months prior to registration
* Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months prior to registration
* Drug induced pneumonitis within 3 months prior to registration
* Signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* Radiographic evidence of cavitating pulmonary lesion(s)
* Tumor invading any major blood vessels
* Evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or mainstem endobronchial tumor within 28 days before the first dose of cabozantinib
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel); allowed anticoagulants are the following:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted
  * Low molecular weight heparins (LMWH) or unfractionated heparin is permitted
  * Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)
* Cardiovascular disorders including:

  * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
  * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days prior to registration
  * Any of the following within 6 months prior to registration:

    * Unstable angina pectoris
    * Clinically-significant cardiac arrhythmias
    * Stroke (including transient ischemic attack [TIA], or other ischemic event)
    * Myocardial infarction
* Gastrointestinal disorders associated with a high risk of perforation or fistula formation within 3 months prior to registration:

  * Active peptic ulcer disease
  * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
  * Known malabsorption syndrome
  * Bowel obstruction or gastric outlet obstruction
  * Percutaneous endoscopic gastrostomy (PEG) tube placement
* Gastrointestinal disorders associated with a high risk of perforation or fistula formation within 6 months prior to registration:

  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess; Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months prior to registration
* Any of the following conditions:

  * Grade 3 or greater infection, or infection requiring intravenous systemic treatment within 28 days prior to registration; patients should be off antibiotics at the time of registration.
  * Serious non-healing wound/ulcer/bone fracture within 28 days prior to registration
  * History of organ transplant
  * Concurrent symptomatic untreated hypothyroidism within 7 days prior to registration
  * History of surgery as follows:

    * Major surgery (as an example, surgery requiring anesthesia and a > 24 hour hospital stay) within 3 months prior to registration, with wound healing at least 28 days prior to registration
    * Minor surgery within 28 days prior to registration with complete wound healing at least 10 days prior to registration
    * Minor procedures within 7 days prior to registration such as thoracentesis, paracentesis, or 18 g or smaller needle biopsy of tumor
    * Patients with clinically relevant ongoing complications from prior surgery are not eligible
* Currently active other malignancies which require systemic treatment
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Active autoimmune disease or known history of autoimmune disease for which recurrence may affect vital organ function or require immune suppressive treatment including systemic corticosteroids; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, autoimmune hepatitis; patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including type I diabetes mellitus or thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Ongoing major illness or psychosocial issues that would limit compliance with the protocol
* Pregnant or breast-feeding
* Patients with known human immunodeficiency virus (HIV) disease taking antiretroviral therapy are excluded because there are no safety data with the combination of antiretroviral therapy and cabozantinib or ipilimumab or nivolumab with ipilimumab

  * Patients with known chronic active hepatitis B (defined as a positive hepatitis B surface antigen and/or hepatitis B viral load in the last

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Neal, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (468):
- United States (468):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on March 1, 2018 and closed on May 31, 2019 for a total of 3 patients enrolled on this study. Patients were randomized to 1 of 3 arms (arms A, B and C). Patients with ROS1 gene rearrangement, MET exon 14 splice mutations, MET high amplification, or RET gene rearrangement were assigned to Arm T.
Period: Overall Study
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib)
Started | 0 | 2 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib) | Total
Number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] |  | 78 [75 to 81] |  | 53 [53 to 53] | 75 [53 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 |  | 1 | 3
  Male |  | 0 |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 |  | 0 | 0
  Not Hispanic or Latino |  | 1 |  | 1 | 2
  Unknown or Not Reported |  | 1 |  | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0 | 0
  Asian |  | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0 | 0
  Black or African American |  | 0 |  | 0 | 0
  White |  | 2 |  | 1 | 3
  More than one race |  | 0 |  | 0 | 0
  Unknown or Not Reported |  | 0 |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as time from randomization to documented disease progression or death from any cause, whichever occurs first. Progression is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions and/or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PFS will be estimated using the Kaplan-Meier method.
Time Frame: Every 3 months up to 4 years and 2 months
Population: All patients enrolled are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib)
Number analyzed (Participants) | 0 | 2 | 0 | 1
months |  | 6.35 [3.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. |  | 14.3 [NA to NA] — Only one patient was enrolled on Arm T so 95% confidence interval was not calculable.

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to death or date last known alive.
Time Frame: Every 3 months up to 4 years and 2 months
Population: All patients enrolled are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib)
Number analyzed (Participants) | 0 | 2 | 0 | 1
months |  | 11.85 [11.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. |  | NA [NA to NA] — The only patient in Arm T was still alive as of the final analysis so median overall survival was not reached and 95% confidence intervals were not calculable.

3. Secondary Outcome: Best Overall Response
Description: Best overall response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Response is defined as either complete response (CR) or partial response (PR).
  Complete response is defined as disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  For Arm T patients, to be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met. Arm A, B, and C patients do not require confirmation scans for CR or PR.
Time Frame: Every 3 months up to 4 years and 2 months
Population: All enrolled patients are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib)
Number analyzed (Participants) | 0 | 2 | 0 | 1
Participants
  Response (CR or PR) |  | 0 |  | 0
  No Response (Other) |  | 2 |  | 1

4. Other Pre Specified Outcome: Progression-free Survival (PFS) by Programmed Death-ligand 1 (PD-L1) Status
Description: as for outcome 1
Time Frame: Every 3 months for 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: The Distribution of Best Overall Response by RECIST 1.1 Criteria, Uni-dimensional Immune Response Criteria (iRRC) and Immune Response Evaluation Criteria in Solid Tumors (iRECIST) Criteria
Description: Best overall response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria:
  Response is defined as either complete response (CR) or partial response (PR). Complete response is defined as disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Response by iRRC is defined as per RECIST1.1.
  Measurements of iRECIST response will be performed as described by Seymour et al with time point and over all response assessments categorized as immune complete response (iCR), immune partial response (iPR), immune stable disease (iSD), immune unconfirmed progressive disease (iUPD) and confirmed progressive disease (iCPD).
Time Frame: Every 3 months for 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Response Per RECIST1.1 Performed by Central Review and by Site Study Personnel
Description: Best overall response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria:
  Response is defined as either complete response (CR) or partial response (PR). Complete response is defined as disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 3 months for 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Effects of Tobacco on Provider-reported Cancer-treatment Toxicity and Dose Modifications
Description: A combined analysis of the data from the selected Eastern Cooperative Oncology Group (ECOG) and the American College of Radiology Imaging Network (ACRIN) trials is planned. Data collected from the tobacco use assessment in each parent study will not be analyzed and reported in the clinical study report.
Time Frame: Assessed every 4 weeks until 30 days after treatment completion, up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Effects of Tobacco on Patient-reported Physical Symptoms and Psychological Symptoms
Description: A combined analysis of the data from the selected ECOG-ACRIN trials is planned. Data collected from the tobacco use assessment in each parent study will not be analyzed and reported in the clinical study report.
  Psychological Symptom Assessment:
  Anxiety & Depression: (The Patient Reported Outcomes Measurement Information System (PROMIS®)). The 4-item Short Form PROMIS® for anxiety and depression will be administered. Score ranges between 4 and 20. Higher scores indicate more anxiety/depression.
  Physical Symptom Assessment by Functional Assessment of Chronic Illness Therapy (FACIT): Six symptom items (general pain, fatigue, nausea, cough, sleep difficulties, shortness of breath) from FACIT will be used for evaluation. Score ranges between 5 and 20. Higher scores indicate higher shame.
Time Frame: Baseline, 3 months and 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assessment of Quitting Behaviors, Behavioral Counseling/Support and Cessation Medication Utilization
Description: A combined analysis of the data from the selected ECOG-ACRIN trials is planned. Data collected from the tobacco use assessment in each parent study will not be analyzed and reported in the clinical study report.
Time Frame: Baseline, 3 months and 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Effects of Tobacco Use and Exposure on Treatment Duration, Relative Dose Intensity, and Therapeutic Benefit
Description: as for outcome 9
Time Frame: Assessed every 3 months for 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 4 years and 2 months
Description: Serious adverse events are defined as grade 3 or higher adverse events that are possibly, probably, or definitely related to protocol therapy. Other adverse events are defined as grade 1 or grade 2 adverse events that are possibly, probably, or definitely related to protocol therapy with a frequency of at least 5% in a given arm.
  All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
Arm/Group | Arm A (Nivolumab) | Arm B (Nivolumab, Cabozantinib) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib)
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/2 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Nivolumab) (N=0) | Arm B (Nivolumab, Cabozantinib) (N=2) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) (N=0) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib) (N=1)
Fatigue (General disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Nivolumab) (N=0) | Arm B (Nivolumab, Cabozantinib) (N=2) | Arm C (Nivolumab, Cabozantinib, Ipilimumab) (N=0) | Arm T (Targeted Cohort; Nivolumab, Cabozantinib) (N=1)
Endocrine disorders - Other, specify (Endocrine disorders) | NA | 1 | NA | 0
Dry eye (Eye disorders) | NA | 1 | NA | 0
Abdominal pain (Gastrointestinal disorders) | NA | 1 | NA | 0
Constipation (Gastrointestinal disorders) | NA | 1 | NA | 0
Diarrhea (Gastrointestinal disorders) | NA | 2 | NA | 0
Dry mouth (Gastrointestinal disorders) | NA | 0 | NA | 1
Mucositis oral (Gastrointestinal disorders) | NA | 1 | NA | 1
Nausea (Gastrointestinal disorders) | NA | 2 | NA | 0
Fatigue (General disorders) | NA | 2 | NA | 0
Autoimmune disorder (Immune system disorders) | NA | 1 | NA | 0
Alanine aminotransferase increased (Investigations) | NA | 2 | NA | 0
Aspartate aminotransferase increased (Investigations) | NA | 1 | NA | 0
Blood bilirubin increased (Investigations) | NA | 2 | NA | 0
Creatinine increased (Investigations) | NA | 1 | NA | 0
Lymphocyte count decreased (Investigations) | NA | 1 | NA | 0
Neutrophil count decreased (Investigations) | NA | 1 | NA | 0
Platelet count decreased (Investigations) | NA | 1 | NA | 0
Weight loss (Investigations) | NA | 1 | NA | 1
White blood cell decreased (Investigations) | NA | 1 | NA | 0
Anorexia (Metabolism and nutrition disorders) | NA | 1 | NA | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | NA | 1 | NA | 0
Hypocalcemia (Metabolism and nutrition disorders) | NA | 1 | NA | 0
Hypophosphatemia (Metabolism and nutrition disorders) | NA | 1 | NA | 0
Dysgeusia (Nervous system disorders) | NA | 1 | NA | 0
Headache (Nervous system disorders) | NA | 1 | NA | 0
Chronic kidney disease (Renal and urinary disorders) | NA | 1 | NA | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | NA | 1 | NA | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03468985/Prot_SAP_000.pdf